CLINICAL TRIAL: NCT02292654
Title: A Phase 1/2, Multi-Center, Open-Label, Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Exploratory Efficacy of Olipudase Alfa in Pediatric Patients Aged <18 Years With Acid Sphingomyelinase Deficiency
Brief Title: Safety, Tolerability, PK, and Efficacy Evaluation of Repeat Ascending Doses of Olipudase Alfa in Pediatric Patients <18 Years of Age With Acid Sphingomyelinase Deficiency
Acronym: ASCEND-Peds
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFI13803; U1111-1160-6469 (Other: UTN)
Record Dates: First submitted 2014-11-07; First posted 2014-11-17 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Sphingomyelin Lipidosis
MeSH Terms: conditions — Niemann-Pick Disease, Type A | interventions — olipudase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olipudase alfa (Experimental): Participants received intravenous (IV) infusion of olipudase alfa once every 2 weeks (Q2W) for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0 milligram per kilogram (mg/kg). Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
  Interventions: Drug: Olipudase alfa

INTERVENTIONS:
Drug: Olipudase alfa — Pharmaceutical form: powder for concentrate for solution for infusion Route of administration: intravenous infusion
  Other Names: GZ402665

SUMMARY:
Primary Objective:

To evaluate the safety and tolerability of olipudase alfa administered intravenously in pediatric participants every 2 weeks for 64 weeks.

Secondary Objective:

To characterize the pharmacokinetic profile and evaluate the pharmacodynamics and exploratory efficacy of olipudase alfa administered intravenously in pediatric participants every 2 weeks for 64 weeks.

DETAILED DESCRIPTION:
The maximum study duration per participant was approximately 18 months (screening period: up to 60 days; treatment period: 64 weeks; post-treatment period: up to 37 days, not applicable if participants enrolled in a long-term extension treatment trial).

ELIGIBILITY:
Inclusion criteria :

* The participant and/or participant's parent(s)/legal guardian(s) must provide written informed assent/consent prior to any protocol-related procedures being performed.
* The participant was <18 years of age on the date of informed assent/consent.
* The participant had documented deficiency of acid sphingomyelinase as measured in peripheral leukocytes, cultured fibroblasts, or lymphocytes.
* The participant had a spleen volume greater than or equal to (>=) 5 multiples of normal (MN) measured by magnetic resonance imaging (MRI); participants who had partial splenectomy were allowed if the procedure was performed >=1 year before screening and the residual spleen volume was >=5 MN.
* The participant's height was -1 Z-score or lower.
* A negative serum pregnancy test in female participants of childbearing potential.
* Female participants of childbearing potential and male participants must be willing to practice true abstinence in line with their preferred and usual lifestyle or use 2 acceptable effective methods of contraception.

Exclusion criteria:

* The participant had received an investigational drug within 30 days before study enrollment.
* The participant had any of the following medical conditions:
* An active, serious, intercurrent illness.
* Active hepatitis B or hepatitis C infection.
* Infection with human immunodeficiency virus (HIV).
* Cirrhosis (determined by clinical evaluation).
* Significant cardiac disease (eg, clinically significant arrhythmia, moderate or severe pulmonary hypertension or valvular dysfunction, or <40 percent (%) left ventricular ejection fraction by echocardiogram).
* Malignancy diagnosed within the previous 5 years (except basal cell carcinoma).
* Any other extenuating circumstance that can significantly interfere with study compliance, including all prescribed evaluations and follow-up activities.
* The participant had acute or rapidly progressive neurological abnormalities.
* The participant was homozygous for SMPD1 gene mutations R496L, L302P, and fs330 or any combination of these 3 mutations.
* The participant had a delay of gross motor skills.
* The participant had a major organ transplant (eg, bone marrow, liver).
* The participant required use of invasive ventilatory support.
* The participant required use of noninvasive ventilatory support while awake and for greater than (>)12 hours a day.
* The participant in the investigator's opinion, was unable to adhere to the requirements of the study.
* The participant had a platelet count <60 × 10^3/µL (based on the average of 2 screening samples obtained up to 24 hours apart).
* The participant had alanine aminotransferase or aspartate aminotransferase >250 IU/L or total bilirubin >1.5 mg/dL.
* The participant had an international normalized ratio (INR) >1.5.
* The participant was unwilling or unable to abstain from ingesting alcohol the day before through 3 days after each infusion of olipudase alfa during the treatment period. Measuring alcohol concentration in blood was not required.
* The participant was scheduled during the study for in-patient hospitalization including elective surgery.
* The participant required medication(s) that may can decrease olipudase alfa activity (eg, fluoxetine, chlorpromazine; tricyclic antidepressants [eg, imipramine, or desipramine]).
* The participant was breast-feeding.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- Investigational Site Number 840001, New York, New York, United States
- Investigational Site Number 076001, Porto Alegre, Brazil
- Investigational Site Number 250002, Bron, France
- Investigational Site Number 276001, Mainz, Germany
- Investigational Site Number 380001, Udine, Italy
- Investigational Site Number 826001, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Diaz GA, Jones SA, Scarpa M, Mengel KE, Giugliani R, Guffon N, Batsu I, Fraser PA, Li J, Zhang Q, Ortemann-Renon C. One-year results of a clinical trial of olipudase alfa enzyme replacement therapy in pediatric patients with acid sphingomyelinase deficiency. Genet Med. 2021 Aug;23(8):1543-1550. doi: 10.1038/s41436-021-01156-3. Epub 2021 Apr 19. PMID 33875845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 sites in 6 countries between 01 May 2015 and 09 December 2019.
Pre-assignment Details: A total of 23 participants were screened out of which 20 participants were included and treated in this study.
Groups:
- Olipudase Alfa: Adolescent Cohort: Participants aged 12 to less than (<) 18 years received intravenous (IV) infusion of olipudase alfa once every 2 weeks (Q2W) for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0 milligram per kilogram (mg/kg). Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
- Olipudase Alfa: Child Cohort: Participants aged 6 to <12 years received IV infusion of olipudase alfa Q2W for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
- Olipudase Alfa: Infant/Early Child Cohort: Participants aged <6 years received IV infusion of olipudase alfa Q2W for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
Period: Overall Study
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Started | 4 | 9 | 7
Completed | 4 | 9 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included all participants who received at least 1 infusion (partial or total) of olipudase alfa.
Groups:
- Olipudase Alfa: Adolescent Cohort: Participants aged 12 to < 18 years received IV infusion of olipudase alfa Q2W for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0 , 3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
- Total: Total of all reporting groups
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total
Number analyzed (Participants) | 4 | 9 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.84 (2.22) | 8.69 (1.69) | 3.77 (1.44) | 8.20 (4.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 4 | 10
  Male | 3 | 4 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Black | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 3 | 7 | 7 | 17
  Southeast Asian | 1 | 1 | 0 | 2
  Northeast Asian | 0 | 0 | 0 | 0
  Not reported | 0 | 0 | 0 | 0
  Other | 0 | 1 | 0 | 1
  Unknown | 0 | 0 | 0 | 0
High Sensitivity C Reactive Protein (hsCRP) Level in Plasma [Mean (Standard Deviation); unit: milligrams per liter (mg/L)] — Population: Here, number analyzed = participants with available data for specified measure.
  milligrams per liter (mg/L)
    number analyzed (Participants) | 4 | 9 | 5 | 18
    (all) | 1.863 (1.855) | 0.410 (0.337) | 0.306 (0.249) | 0.704 (1.041)
Safety Biomarker: Ceramide Level in Plasma [Mean (Standard Deviation); unit: mg/L] | 7.13 (2.14) | 5.57 (1.87) | 8.01 (5.30) | 6.74 (3.51)
Safety Biomarker: Iron Level in Plasma [Mean (Standard Deviation); unit: micromole/liter (umol/L)] — Population: Here, number analyzed = participants with available data for specified measure.
  micromole/liter (umol/L)
    number analyzed (Participants) | 4 | 9 | 5 | 18
    (all) | 10.13 (2.38) | 10.96 (2.31) | 8.52 (1.81) | 10.09 (2.32)
Safety Biomarker: Cardiac Troponin I Level in Plasma [Mean (Standard Deviation); unit: micrograms per liter (μg/L)] — Population: Here, number analyzed = participants with available data for specified measure.
  micrograms per liter (μg/L)
    number analyzed (Participants) | 4 | 9 | 5 | 18
    (all) | 0.020 (0.000) | 0.020 (0.000) | 0.020 (0.000) | 0.020 (0.000)
Safety Biomarker: Ferritin Level in Plasma [Mean (Standard Deviation); unit: μg/L] | 65.775 (21.088) | 68.700 (36.733) | 46.329 (26.500) | 60.285 (31.173)
Safety Biomarker: Interleukin (IL)-6 Level in Plasma [Mean (Standard Deviation); unit: nanogram/liter (ng/L)] — Population: Here, number analyzed = participants with available data for specified measure. Here, number analyzed = '0' represented that data were not calculated for specified category due to non-availability of evaluable participants.
  nanogram/liter (ng/L)
    number analyzed (Participants) | 4 | 9 | 0 | 13
    (all) | 2.27 (0.87) | 11.15 (25.62) |  | 8.73 (21.84)
Safety Biomarker: IL-8 Level in Plasma [Mean (Standard Deviation); unit: ng/L] — Population: Here, number analyzed = participants with available data for specified measure. Here, number analyzed = '0' represented that data were not calculated for specified category due to non-availability of evaluable participants.
  ng/L
    number analyzed (Participants) | 4 | 9 | 0 | 13
    (all) | 24.75 (14.50) | 35.72 (29.15) |  | 32.35 (25.43)
Safety Biomarker: Calcitonin Level in Plasma [Mean (Standard Deviation); unit: ng/L] | 7.675 (13.330) | 9.031 (8.601) | 12.991 (7.843) | 10.146 (9.137)
Percent Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: percent ejection fraction] — Population: Here, number analyzed = participants with available data for specified measure.
  percent ejection fraction
    number analyzed (Participants) | 4 | 8 | 7 | 19
    (all) | 60.50 (4.04) | 64.25 (6.27) | 68.71 (7.16) | 65.11 (6.72)
Pharmacodynamic Biomarker: Sphingomyelin in Plasma [Mean (Standard Deviation); unit: mg/L] | 348.3 (27.5) | 430.8 (191.3) | 318.7 (41.0) | 375.1 (137.3)
Pharmacodynamic Biomarker: Lyso-Sphingomyelin in Plasma [Mean (Standard Deviation); unit: ug/L] | 488.250 (153.489) | 653.667 (226.301) | 670.000 (382.137) | 626.300 (276.528)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) that occurred or worsened during the on-treatment period (time from the start of investigational medicinal product [IMP]) administration until end of study (i.e. up to 64 weeks).
Time Frame: From Baseline up to End of study (64 weeks)
Population: Safety population included all participants who received at least 1 infusion (partial or total) of olipudase alfa.
Measure: Count of Participants; unit: Participants
Groups:
- Olipudase Alfa: Adolescent Cohort: Participants aged 12 to <18 years received IV infusion of olipudase alfa Q2W for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0 , 3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
- Total Participants: All participants received IV infusion of olipudase alfa Q2W for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0 mg/kg. The target maintenance dose was 3.0 mg/kg, which was maintained for the remaining duration of 64 treatment weeks.
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants
  Any TEAEs | 4 | 9 | 7 | 20
  Any TEAEs leading to death | 0 | 0 | 0 | 0
  Any TEAEs leading to dose reduction | 0 | 4 | 3 | 7
  Any TEAEs potentially related to study drug | 2 | 6 | 5 | 13

2. Primary Outcome: Number of Participants With Infusion-Associated Reactions (IARs)
Description: IARs were defined as AEs that occurred during the infusion or within up to 24 hours after the start of infusion and were considered as related or possibly related to the study treatment by the investigator or the sponsor. Protocol-defined IAR: all AEs that were identified as an IAR by the investigator. Events occurring greater than or equal to (>=) 24 hours after the start of an infusion might had been judged an IAR at the discretion of the investigator or sponsor.
Time Frame: Within up to 24 hours after start of any infusion (during the treatment period i.e. from Baseline up to 64 weeks)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Groups:
- Olipudase Alfa: Adolescent Cohort: Participants aged 12 to <18 years received IV infusion of olipudase alfa Q2W for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3,0.3, 0.6, 0.6, 1.0, 2.0 , 3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants | 0 | 6 | 5 | 11

3. Primary Outcome: Number of Participants With Change in Physical Examination
Description: Change from Normal assessment (at Baseline) to Abnormal assessment (at Week 52) was reported. Physical examinations included following observations/measurements: examination of the skin, head, eyes, ears, nose, and throat; lymph nodes; heart, lungs, and abdomen; extremities and joints. Abnormality in physical examinations was based on investigator's discretion.
Time Frame: Baseline, Week 52 (last complete assessment)
Population: Analysis was performed on safety population. One participant may be counted in multiple categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants
  Abdomen | 0 | 0 | 0 | 0
  Heart | 0 | 0 | 0 | 0
  Skin | 0 | 1 | 1 | 2
  Extremities/Joints | 0 | 1 | 0 | 1
  General Appearance | 0 | 1 | 1 | 2
  Head, Eyes, Ears, Nose and Throat | 2 | 0 | 2 | 4
  Lymph Nodes | 0 | 0 | 0 | 0
  Lungs | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Change in Neurological Examination
Description: Change from Normal assessment (at Baseline) to Abnormal assessment (at Week 52) was reported. Neurological examination included: coordination examination, cranial nerve examination, extrapyramidal features, fundoscopy, gait and coordination examination, motor examination, tone peripheral nervous system, reflexes examination, sensory examination, strength examination, mental status.
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis was performed on safety population. One participant may be counted in multiple categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants
  Coordination Examination | 0 | 0 | 0 | 0
  Cranial Nerve Examination | 0 | 0 | 0 | 0
  Extrapyramidal Features | 0 | 0 | 0 | 0
  Fundoscopy | 0 | 0 | 1 | 1
  Gait and Coordination Examination | 0 | 0 | 0 | 0
  Motor Examination, Tone | 0 | 0 | 0 | 0
  Peripheral Nervous System | 0 | 0 | 0 | 0
  Reflexes Examination | 0 | 0 | 0 | 0
  Sensory Examination | 0 | 0 | 0 | 0
  Strength Examination | 0 | 0 | 1 | 1
  Mental Status | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Liver Function Laboratory Values at the End of Study
Description: Abnormal values in alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, and alkaline phosphatase were reported.
Time Frame: At End of Study (Week 64)
Population: Analysis was performed on safety population. One participant may be counted in multiple categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants
  ALT | 0 | 1 | 1 | 2
  AST | 0 | 1 | 0 | 1
  Total Bilirubin | 0 | 0 | 0 | 0
  Alkaline Phosphatase | 2 | 2 | 0 | 4

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Abnormalities
Description: * Heart Rate (HR) High: >=120 beats per minute (bpm) (adolescents), >=120 bpm (children), >=140 bpm (early children), >=175 bpm (infants) & increase from baseline (IFB) >=20 bpm for all age categories.
  * HR Low: <=50 bpm (adolescents), <=50 bpm (children), <=75 bpm (early children), <=80 bpm (infants) & decrease from baseline (DFB) >=20 bpm for all age categories.
  * Systolic BP (SBP) High: >=119 mmHg (adolescents), 108 mmHg (children), 101 mmHg (in early children), 98 mmHg (infants) & IFB >=20 mmHg for all age categories.
  * SBP Low: <=90 mmHg (adolescents), <= 80mm Hg (children), <=70 mmHg (early children), <=70 mmHg (infants) & DFB >=20 mmHg for all age categories.
  * Diastolic BP (DBP) High:>=78 mmHg (adolescents), >=72 mmHg (children), >=59 mmHg (in early children), >=54 mmHg (infants) & IFB >=10 mmHg for all age categories.
  * DBP Low:<=54 mmHg (adolescents), <=48 mmHg (children), <=34 mmHg (early children), <=34 mmHg (infants) & DFB >=10 mmHg for all age categories.
Time Frame: From Baseline up to End of Study (64 weeks)
Population: Analysis was performed on safety population. One participant may be counted in multiple (more than 1) categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants
  Heart Rate High | 0 | 5 | 3 | 8
  Heart Rate Low | 1 | 0 | 7 | 8
  SBP High | 3 | 6 | 6 | 15
  SBP Low | 2 | 5 | 0 | 7
  DBP High | 4 | 8 | 7 | 19
  DBP Low | 4 | 9 | 2 | 15

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for potentially clinically significant ECG abnormalities:
  * High PR Interval: >=180 milliseconds (ms) in adolescents, 170 ms in children, 160 ms in early children, and 140 ms in infants;
  * High QRS Interval: >=110 ms in adolescents, 100 ms in children, 95 ms in early children and 85 ms in infants;
  * Prolonged QTc Fridericia (QTc F): >450 ms in male adolescents, children, early children and infants or 470 ms in female adolescents,
  * QTc F >500 ms;
  * QTc F increase from baseline >60 ms.
Time Frame: From Baseline up to End of Study (64 weeks)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants
  High PR Duration | 2 | 2 | 2 | 6
  High QRS Duration | 0 | 0 | 0 | 0
  Prolonged QTc F | 1 | 1 | 0 | 2
  QTc F >500 ms | 0 | 0 | 0 | 0
  QTc F increase from baseline >60 ms | 0 | 0 | 0 | 0

8. Primary Outcome: Change From Baseline in Safety Biomarker Level: High Sensitivity C Reactive Protein (hsCRP) at Week 64
Time Frame: Baseline, Week 64 (pre-infusion)
Population: Analysis was performed on safety population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 5 | 18
mg/L | -1.603 (1.976) | -0.168 (0.411) | -0.206 (0.249) | -0.497 (1.074)

9. Primary Outcome: Change From Baseline in Safety Biomarker: Ceramide Level at Week 64
Time Frame: Baseline, Week 64 (pre-infusion)
Population: Analysis was performed on safety population.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Olipudase Alfa: Adolescent Cohort: Participants aged 12 to <18 years received IV infusion of olipudase alfa Q2W for 64 weeks. Each participant underwent a dose escalation according to the following paradigm: 0.03, 0.1, 0.3, 0.3, 0.6, 0.6, 1.0, 2.0, 3.0 mg/kg. Three (3) mg/kg was the target maintenance dose, which was maintained for the remaining duration of 64 treatment weeks.
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
mg/L | -3.90 (2.41) | -3.23 (2.17) | -5.93 (4.91) | -4.31 (3.48)

10. Primary Outcome: Change From Baseline in Safety Biomarker: Iron at Week 64
Time Frame: Baseline, Week 64 (pre-infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 8 | 5 | 17
umol/L | 1.40 (3.53) | -0.41 (5.07) | 1.52 (4.31) | 0.58 (4.38)

11. Primary Outcome: Change From Baseline in Safety Biomarker: Cardiac Troponin I and Ferritin at Week 64
Time Frame: Baseline, Week 64 (pre-infusion)
Population: Analysis was performed on safety population. Here 'number analyzed' = participants with available data for specified categories.
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
μg/L
  Troponin: Pre-infusion: Week 64: number analyzed (Participants) | 4 | 9 | 5 | 18
  Troponin: Pre-infusion: Week 64 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  Ferritin: Pre-infusion: Week 64 | -38.325 (16.438) | -45.611 (32.963) | -28.186 (19.793) | -38.055 (26.207)

12. Primary Outcome: Change From Baseline in Safety Biomarker: Interleukin (IL)-6 and IL-8 at Week 24
Time Frame: Baseline, Week 24 (pre-infusion, last assessment)
Population: Analysis was performed on safety population. Here 'number analyzed'=participants with available data for specified categories. Data was not planned to be collected and reported for the Infant/Early Child Cohort, per protocol.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 13
ng/L
  IL-6: number analyzed (Participants) | 3 | 8 | 11
  IL-6 | 0.47 (3.23) | 0.89 (5.66) | 0.77 (4.95)
  IL-8 | -7.25 (14.50) | -18.22 (29.15) | -14.85 (25.43)

13. Primary Outcome: Change From Baseline in Safety Biomarker: Calcitonin at Week 64
Time Frame: Baseline, Week 64 (pre-infusion)
Population: Analysis was performed on safety population.
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
ng/L | 3.612 (7.225) | -5.337 (3.962) | -8.609 (6.359) | -4.710 (6.929)

14. Primary Outcome: Doppler Echocardiogram: Absolute Change From Baseline in Left Ventricular Ejection Fraction at Week 52
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 3 | 7 | 6 | 16
percent ejection fraction | 0.33 (4.51) | -1.00 (5.16) | 1.17 (4.83) | 0.06 (4.71)

15. Primary Outcome: Number of Participants With Treatment-Emergent Antibody: Treatment-Induced/Treatment-Boosted Anti-drug Antibodies and Neutralizing Antibody (NAb)
Description: Serum samples for immunogenicity assessment were analyzed to detect ADA. ADA response were categorized as: treatment emergent antibody i.e. treatment-induced/treatment-boosted response. A participant whose ADA status was positive anytime post-baseline and was negative or missing at baseline was considered to have treatment induced ADA. A participant whose ADA status was positive at baseline (pre-existing ADA) and the ADA titer level anytime post-baseline was significantly higher than that at baseline is considered to have treatment boosted ADA. Positive samples in the ADA assay were further analyzed in the NAb assay as positive NAb inhibition of catalytic activity and positive NAb inhibition of cellular uptake.
Time Frame: From Baseline up to Week 64
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants
  ADA positive since first dose of olipudase alfa | 2 | 7 | 3 | 12
  Positive NAb of catalytic activity | 0 | 1 | 0 | 1
  Positive NAb of cellular uptake | 0 | 0 | 0 | 0
  Treatment Induced ADA | 2 | 6 | 3 | 11
  Treatment boosted ADA | 0 | 1 | 0 | 1

16. Primary Outcome: Number of Participants With Abnormalities in Liver Ultrasound Doppler at Week 52
Description: Evidence of portal hypertension was assessed by portal vein direction from liver ultrasound doppler.
Time Frame: Week 52 (last assessment)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
Participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Pharmacokinetic (PK) Parameter: Plasma Concentration of Olipudase Alfa at the End of Infusion (Ceoi)
Description: Ceoi was defined as the plasma concentration at the end of infusion (EOI). Data collected for child and Infant/child age groups at 0-30 min from end of infusion was considered at end of infusion.
Time Frame: At the end of infusion of the first 3.0 mg/kg dose and at Week 52
Population: Analysis was performed on PK population which included all participants who received at least 1 infusion of study medication and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Number analyzed (Participants) | 4 | 9 | 7
micrograms per milliliter (μg/mL)
  3.0 mg/kg at First dose | 28.0 (4.88) | 23.0 (3.93) | 22.1 (7.19)
  3.0 mg/kg at Day 52 | 22.4 (1.02) | 24.4 (7.51) | 22.4 (4.18)

18. Secondary Outcome: Pharmacokinetic Parameter: Maximum Observed Plasma Concentration (Cmax) of Olipudase Alfa
Description: Cmax: maximum plasma concentration observed.
Time Frame: Adolescent: at pre-infusion, EOI, 2 h, 6 h, 24 h, 48 h & 72 h (at first 3.0 mg/kg dose) or 96 h (at Week 52) post EOI; Child & infant/early child: pre-infusion, 0-30 min, 2-4 h, 6-12 h, 24-36 h, and 84-96 h post EOI at the first 3.0 mg/kg dose & Week 52
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Number analyzed (Participants) | 4 | 9 | 7
μg/mL
  3.0 mg/kg at First dose | 28.0 (4.88) | 23.0 (3.93) | 22.1 (7.19)
  3.0 mg/kg at Week 52 | 22.4 (1.02) | 24.4 (7.51) | 22.4 (4.18)

19. Secondary Outcome: Pharmacokinetic Parameter: AUC0-last, AUC(0-tau) of Olipudase Alfa
Description: AUClast: Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the time of last measured concentration.
  AUC(0-tau): area under the plot of the drug concentration versus the time curve from time "0" to the end of the dosing interval (tau), where dosing interval was 2 weeks.
Time Frame: as for outcome 18
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: μg*h/mL
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Number analyzed (Participants) | 4 | 9 | 7
μg*h/mL
  AUClast: at 3.0 mg/kg First dose | 452 (49.7) | 441 (97.8) | 412 (87.4)
  AUClast: at 3.0 mg/kg at Week 52 | 461 (28.1) | 482 (101) | 429 (62.6)
  AUC(0-τ): at 3.0 mg/kg First dose | 478 (55.4) | 465 (102) | 432 (93.0)
  AUC(0-τ): at 3.0 mg/kg at Week 52 | 489 (32.7) | 508 (108) | 451 (68.2)

20. Secondary Outcome: Pharmacokinetic Parameter: Terminal Half-Life of Olipudase Alfa
Description: Half-life is the time measured for the plasma concentration of drug to decrease by one half.
Time Frame: as for outcome 18
Population: Analysis was performed on PK population
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Number analyzed (Participants) | 4 | 9 | 7
hours (h)
  3.0 mg/kg at First dose | 17.1 (1.15) | 23.1 (2.11) | 22.6 (1.25)
  3.0 mg/kg at Week 52 | 24.3 (2.88) | 23.3 (1.42) | 23.6 (1.35)

21. Secondary Outcome: Pharmacokinetic Parameter: Total Body Clearance (CL) of Olipudase Alfa
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Total body clearance of a drug from the plasma calculated using equations below: CL = Dose / AUC after the first dose.
Time Frame: as for outcome 18
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: milliliter/hour/kilograms (mL/h/kg)
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Number analyzed (Participants) | 4 | 9 | 7
milliliter/hour/kilograms (mL/h/kg)
  3.0 mg/kg at First dose | 6.34 (0.741) | 6.75 (1.57) | 7.20 (1.40)
  3.0 mg/kg at Week 52 | 6.16 (0.411) | 6.16 (1.38) | 6.79 (1.08)

22. Secondary Outcome: Pharmacokinetic Parameter: Volume of Distribution at Steady State (Vss) of Olipudase Alfa
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: as for outcome 18
Population: Analysis was performed on PK population.
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Number analyzed (Participants) | 4 | 9 | 7
milliliter per kilogram (mL/kg)
  3.0 mg/kg at First dose | 133 (13.5) | 166 (39.1) | 165 (31.0)
  3.0 mg/kg at Week 52 | 172 (11.6) | 153 (32.7) | 161 (20.9)

23. Secondary Outcome: Pharmacokinetic Parameter: Time to Reach Cmax (Tmax) of Olipudase Alfa
Description: tmax: time to reach maximum plasma concentration observed.
Time Frame: as for outcome 18
Population: Analysis was performed on PK population.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort
Number analyzed (Participants) | 4 | 9 | 7
hours (h)
  3.0 mg/kg at First dose | 3.94 [3.87 to 4.08] | 4.00 [3.83 to 7.07] | 4.13 [3.75 to 8.70]
  3.0 mg/kg at Week 52 | 3.81 [3.67 to 4.03] | 4.25 [3.75 to 9.78] | 4.42 [4.08 to 5.87]

24. Secondary Outcome: Percent Change From Baseline in Spleen Volume and Liver Volume at Week 52
Description: Spleen and liver volumes was assessed by abdominal magnetic resonance imaging (MRI).
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all participants who were exposed to IMP, regardless of the amount of treatment administered (partial or total).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
percent change
  Change in spleen volume | -46.936 (3.041) | -46.038 (11.767) | -54.590 (7.562) | -49.211 (9.713)
  Change in liver volume | -41.726 (6.130) | -36.741 (10.469) | -45.060 (8.203) | -40.560 (9.370)

25. Secondary Outcome: Change From Baseline in Interstitial Lung Disease Score Measured Using High Resolution Computed Tomography (HRCT) at Week 52 For Both Lungs
Description: Pulmonary imaging of chest using HRCT was obtained to quantitate the degree of possible infiltrative lung disease. Lung fields were assessed by a central reader & scored subjectively for the degree of interstitial lung disease on a scale ranges from 0 =normal, 1 =mild, 2=moderate and 3 =severe, where higher scores indicate more severity.
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 6 | 19
score on a scale | -0.2188 (1.0020) | -0.5833 (0.7906) | -0.8958 (0.9982) | -0.6053 (0.8851)

26. Secondary Outcome: Change From Baseline in Height Z-Scores at Week 52
Description: Z-score for height of participants was evaluated. Height Z-Score, i.e., the height-for-age Z Score, is the number of standard deviations of the actual height of a child from the median height of the children of the corresponding age and sex as determined from the standard sample. A height Z-score of 0 is equal to the median and is considered normal. Negative numbers indicate values lower than the median and positive numbers indicate values higher than the median. For analysis, mean Z-score was calculated and an increase of mean height Z-score from baseline indicates an improvement on growth.
Time Frame: Baseline, Week 52 (last assessment)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 8 | 7 | 19
Z-score | 0.606 (0.290) | 0.371 (0.344) | 0.736 (0.423) | 0.555 (0.385)

27. Secondary Outcome: Percent Change From Baseline in Percent Predicted Hemoglobin-Adjusted Diffusing Capacity of Carbon Monoxide (DLco) at Week 52
Description: Percent predicted Hemoglobin-adjusted DLco was calculated as: 100*Adjusted DLco/Predicted DLco in unit of mL CO/min/mmHg where, adjusted DLco = Observed DLco (in mL CO/min/mmHg) divided by Hemoglobin-adjusted factor. Per planned analysis, pulmonary function testing (PFT) was to be performed only on participants >=5 years of age therefore, data for participants in "age cohort: infant/early child" were not collected.
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis was performed on mITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure. PFT was to be performed only on participants >=5 years of age and who could perform the test, therefore, for participants in "age cohort: infant/early child" data were not collected.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort
Number analyzed (Participants) | 3 | 6
percent change | 28.01 (16.22) | 35.41 (35.08)

28. Secondary Outcome: Change From Baseline in Difference Between Actual Age and Bone Age of Participants at Week 52
Description: Hand X-ray was performed on participant's left hand, fingers and wrist to assess bone age of participants. At each visit (Baseline and Week 52), difference between the bone age and actual age at that visit was calculated. Difference in age in months was calculated as bone age in months minus real age at time of assessment (in months) at specified time points. In this outcome measure change from baseline at Week 52 in the difference between actual age and bone age (in months) is reported.
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
months | 1.595 (3.114) | 2.876 (14.048) | -0.702 (9.573) | 1.368 (10.781)

29. Secondary Outcome: Change From Baseline in Cycle Ergometry: Maximum Workload at Week 52
Description: Cardiopulmonary status was assessed using a stationary one-wheeled cycle used as an ergometer to measure a person's work output under controlled conditions. Participants were asked to ride the cycle at increasing workload levels until they could no longer proceed. The workload at which participant stopped and cannot proceed was considered as maximum workload (in watt). As per the planned analysis, this assessment was not to be performed on participants that were <=6 years of age or <120 cm in height on day 1/week 0, therefore infant/early child cohort was not evaluable.
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis was performed on mITT population. Here, overall number of participants analysed = participants with available data for this outcome measure. Data not collected in participants <=6 years old, per protocol.
Measure: Mean (Standard Deviation); unit: watts
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort
Number analyzed (Participants) | 3 | 2
watts | 38.3 (10.7) | 20.5 (7.8)

30. Secondary Outcome: Physician's Global Assessment of Participant's Progress: Observed Scores at Week 52
Description: Physician assessed participant's current clinical status (refers to clinical status at Week 52 in comparison to Baseline) was evaluated by marking 1 of the following 7 categories: • marked improvement, • moderate improvement, • mild improvement, • no change, • mild worsening, • moderate worsening, or • marked worsening. These 7 categories were converted to scores as follows: 3 = marked improvement of daily activities, 2 = moderate improvement of daily activities, 1 = mild improvement of daily activities, 0 = no change, -1 = mild worsening of daily activities, -2 = moderate worsening of daily activities, -3 = marked worsening of daily activities where higher score indicated improvement in daily activities as compared to baseline. In this outcome measure, observed scores of participant's clinical status at Week 52 are reported.
Time Frame: Week 52 (last assessment)
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
score on a scale | 1.3 (1.5) | 2.4 (1.0) | 2.7 (0.8) | 2.3 (1.1)

31. Secondary Outcome: Percent Change From Baseline in Efficacy Biomarkers Level at Week 52
Description: Efficacy biomarkers included chitotriosidase, chemokine ligand 18 (CCL18), angiotensin-converting enzyme (ACE).
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population. Here 'number analyzed' = participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
percent change
  Chitotriosidase at Week 52: number analyzed (Participants) | 4 | 8 | 7 | 19
  Chitotriosidase at Week 52 | -55.8 (21.1) | -44.7 (25.0) | -74.6 (18.1) | -58.0 (24.8)
  CCL18 at Week 52 | -55.25 (13.23) | -66.20 (22.97) | -68.13 (16.63) | -64.68 (19.01)
  ACE at Week 52 | -29.92 (19.59) | -24.57 (14.15) | -29.64 (17.80) | -27.41 (15.87)

32. Secondary Outcome: Percent Change From Baseline in Lipid Profile at Week 52
Description: Lipid profile parameters included low density lipoprotein (LDL)-cholesterol, high density lipoprotein (HDL)-cholesterol and triglycerides.
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for specified category.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
percent change
  LDL Cholesterol at Week 52: number analyzed (Participants) | 4 | 9 | 6 | 19
  LDL Cholesterol at Week 52 | -38.31 (7.44) | -35.82 (23.00) | -34.04 (16.69) | -35.78 (18.00)
  HDL Cholesterol at Week 52 | 118.63 (66.75) | 87.49 (52.89) | 124.74 (84.57) | 106.76 (66.82)
  Triglycerides at Week 52 | -56.28 (5.95) | -47.45 (18.08) | -56.44 (25.01) | -52.37 (19.02)

33. Secondary Outcome: Percent Change From Baseline in Bone Biomarkers at Week 52
Description: Bone biomarkers included bone specific alkaline phosphatase, C-Telopeptide.
Time Frame: Baseline, Week 52
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
percent change
  Alkaline phosphatase: Week 52: number analyzed (Participants) | 3 | 9 | 5 | 17
  Alkaline phosphatase: Week 52 | -9.154 (50.568) | 44.768 (50.111) | 35.040 (61.983) | 32.391 (54.292)
  C-Telopeptide: Week 52: number analyzed (Participants) | 4 | 8 | 5 | 17
  C-Telopeptide: Week 52 | 69.0 (93.7) | 92.5 (78.4) | 50.6 (37.0) | 74.7 (70.9)

34. Secondary Outcome: Change From Baseline in Health Outcome Questionnaires : Pediatric Quality of Life (PedsQL) Generic Core Total Scale Scores at Week 52
Description: PedsQL includes a child self-report (CS-R) for participants 5 to 18 years and parents' report (PR) of participants 2 to 18 years. CS-R: 23-item PedsQL Generic Core Scales report includes 4 scales, Physical (P), Emotional (E), Social (S), and School Functioning (SF). PR: 21-item PedsQL Generic Core Scales report includes P, E, S, and SF scales. Each item used a 5-point rating scale ( from 0=never to 4=almost always). Items are reverse scored and linearly transformed to a 0 (almost always) -100 (never) scale. Higher score indicates better Health Related Quality of Life (HRQoL). P, E, S and SF summary scores are calculated as mean of respective functioning items. Psychosocial Health Summary Score is calculated as mean of 13 or 15 items (E, S and SF). Generic core total scale score is calculated as the mean of all the 21 or 23 items (P, E, S and SF). All summary/total scores are mean of specific items and they all have values ranges from 0 to 100, where higher score=better HRQoL.
Time Frame: Baseline, Week 52 (last assessment)
Population: Analysis performed on mITT population. Number of participants analyzed=participants with available data. PedsQL includes CS-R age 5 to18 (scoring categories 5 to 7, 8 to 12 and 13 to 18 years); PR age 2 to 18 (scoring categories 2 to 4, 5 to 7, 8 to 12 and 13 to 18 years). Since PedsQL scoring age categories are not the same as the age cohort defined for the study and since this is a single arm study, overall mITT population with available data is reported for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Total Participants
Number analyzed (Participants) | 19
score on a scale
  Physical Functioning Scale: Child Report: number analyzed (Participants) | 13
  Physical Functioning Scale: Child Report | 9.4 (7.9)
  Emotional Functioning Scale: Child Report: number analyzed (Participants) | 13
  Emotional Functioning Scale: Child Report | 14.6 (15.1)
  Social Functioning Scale: Child Report: number analyzed (Participants) | 13
  Social Functioning Scale: Child Report | 4.2 (13.2)
  School Functioning Scale: Child Report: number analyzed (Participants) | 13
  School Functioning Scale: Child Report | 2.1 (12.6)
  Psychosocial Health Summary Score: Child Report: number analyzed (Participants) | 13
  Psychosocial Health Summary Score: Child Report | 6.8 (8.3)
  Generic Core Total Scale Score : Child Report: number analyzed (Participants) | 13
  Generic Core Total Scale Score : Child Report | 7.6 (5.5)
  Physical Functioning Scale: Parent Report: number analyzed (Participants) | 18
  Physical Functioning Scale: Parent Report | 15.5 (15.3)
  Emotional Functioning Scale: Parent Report: number analyzed (Participants) | 18
  Emotional Functioning Scale: Parent Report | 12.2 (22.9)
  Social Functioning Scale:Parent Report: number analyzed (Participants) | 18
  Social Functioning Scale:Parent Report | 11.7 (19.8)
  School Functioning Scale: Parent Report: number analyzed (Participants) | 17
  School Functioning Scale: Parent Report | 1.0 (20.5)
  Psychosocial Health Summary Score:Parent Report: number analyzed (Participants) | 18
  Psychosocial Health Summary Score:Parent Report | 8.2 (14.5)
  Generic Core Total Scale Score: Parent Report: number analyzed (Participants) | 18
  Generic Core Total Scale Score: Parent Report | 10.8 (13.4)

35. Secondary Outcome: Percent Change From Baseline in Pharmacodynamic Biomarkers: Plasma Sphingomyelin and Lyso-Sphingomyelin Levels at Week 52
Description: Sphingomyelin and Lyso-sphingomyelin levels were assessed in plasma. Lyso-sphingomyelin is a metabolite of sphingomyelin.
Time Frame: Baseline, Week 52 (Pre- infusion)
Population: Analysis was performed on PD population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
Number analyzed (Participants) | 4 | 9 | 7 | 20
percent change
  Sphingomyelin: Pre-infusion at Week 52 | -4.4 (24.6) | -37.1 (24.2) | -18.6 (40.3) | -24.1 (32.0)
  Lyso-Sphingomyelin: Pre-infusion at Week 52 | -84.050 (5.249) | -88.029 (8.156) | -87.951 (1.775) | -87.206 (5.998)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from first IMP administration up to 64 weeks regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that is AEs that developed/worsened during the 'on-treatment period' (time from the start of first infusion until 64 weeks). The other Non-serious adverse events section contains Events >=2% and participants >=2. Analysis was performed on safety population.
Arm/Group | Olipudase Alfa: Adolescent Cohort | Olipudase Alfa: Child Cohort | Olipudase Alfa: Infant/Early Child Cohort | Total Participants
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9 | 0/7 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/9 | 4/7 | 5/20
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9 | 7/7 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olipudase Alfa: Adolescent Cohort (N=4) | Olipudase Alfa: Child Cohort (N=9) | Olipudase Alfa: Infant/Early Child Cohort (N=7) | Total Participants (N=20)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pneumonia Mycoplasmal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (3) | 1 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olipudase Alfa: Adolescent Cohort (N=4) | Olipudase Alfa: Child Cohort (N=9) | Olipudase Alfa: Infant/Early Child Cohort (N=7) | Total Participants (N=20)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 5 (19) | 1 (1) | 6 (20)
Diarrhoea (Gastrointestinal disorders) | 2 (5) | 5 (10) | 4 (7) | 11 (22)
Vomiting (Gastrointestinal disorders) | 2 (3) | 6 (21) | 4 (14) | 12 (38)
Pyrexia (General disorders) | 1 (3) | 7 (24) | 7 (29) | 15 (56)
Nasopharyngitis (Infections and infestations) | 2 (4) | 5 (13) | 4 (11) | 11 (28)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (4) | 5 (13) | 8 (17)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (55) | 3 (33) | 6 (88)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 2 (36) | 2 (8) | 4 (44)
Headache (Nervous system disorders) | 2 (12) | 5 (21) | 1 (5) | 8 (38)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 7 (15) | 5 (13) | 14 (31)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6) | 1 (11) | 4 (17)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (5) | 3 (13) | 6 (18)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (13) | 2 (3) | 5 (16)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (20) | 1 (3) | 3 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT02292654/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT02292654/SAP_001.pdf